CLINICAL TRIAL: NCT06219369
Title: Comparison of Postoperative Analgesic Efficacy of Serratus Posterior Superior Intercostal Plane Block and Thoracic Paravertebral Block in Patients Undergoing Video-Assisted Thoracoscopic Surgery
Brief Title: Effecot of Serratus Posterior Superior Intercostal Plane Block and Thoracic Paravertebral Block in VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Collaborators: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Güvenç Doğan, Associate Professor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hitit
Record Dates: First submitted 2023-12-29; First posted 2024-01-23 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Video-assisted Thoracoscopic Surgery
Keywords: thoracic paravertebral block; VATS; serratus posterior superior interkostal plane block
MeSH Terms: interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: SPSIPB Technique:
  The SPSIPB block, which follows the guidelines we routinely use, will be performed after the completion of the surgical procedure and before the patient wakes up.
  TPVB Technique:
  The US probe (11-12 MHz, Vivid Q) will be placed 2-3 cm lateral to the T5 spinous process. After visualizing the transverse process, the paravertebral area, internal intercostal membrane, paravertebral space, and pleura, the needle will be advanced to the paravertebral space using an in-plane technique.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Active Comparator): Group T patients who underwent TPVB
  Interventions: Procedure: Group T
- Group S (Active Comparator): Group S patients who underwent SPSIPB
  Interventions: Procedure: Group T

INTERVENTIONS:
Procedure: Group T — SPSIPB Technique:
  The SPSIPB block, which follows the guidelines we routinely use, will be performed after the completion of the surgical procedure and before the patient wakes up.
  TPVB Technique:
  The US probe (11-12 MHz, Vivid Q) will be placed 2-3 cm lateral to the T5 spinous process. After visualizing the transverse process, the paravertebral area, internal intercostal membrane, paravertebral space, and pleura, the needle will be advanced to the paravertebral space using an in-plane technique.
  Other Names: Group S

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) has become a standard procedure in both minor and major lung surgeries in thoracic surgery operations. Although postoperative pain in patients undergoing VATS is not as severe as that seen after thoracotomy, it still occurs. This, in turn, affects postoperative pulmonary complications and patients' lengths of hospital stay. Thoracic epidural analgesia (TEA) is still considered the gold standard in the treatment of postoperative pain. However, due to side effects such as post-procedural hypotension, urinary retention, or nausea/vomiting, alternative analgesic methods such as thoracic paravertebral block (TPVB), intercostal block, serratus anterior plane block (SAPB), erector spinae plane block (ESPB), and serratus posterior superior intercostal plane block (SPSIPB) are being considered instead of epidural analgesia.

Among these methods, TPVB performed under ultrasound guidance is already a commonly preferred and classical method. In patients undergoing thoracotomy and VATS, Tulgar and colleagues have defined SPSIPB as a new technique and demonstrated its efficacy in providing analgesia in the hemithorax when considering the sensory dermatome of SPSIPB in a cadaveric and a case series study with five patients conducted in 2023. Similarly, Avcı and colleagues, in their article published in 2023, emphasized the analgesic effectiveness of SPSIPB in the thoracic region after VATS. As far as we know, there is no published study comparing TPVB and SPSIPB under ultrasound guidance to date. Therefore, the aim of this study was to compare ultrasound-guided TPVB and SPSIPB in postoperative analgesia after VATS. Our primary goal is to investigate whether there are any superiority in terms of postoperative Visual analog score (VAS), time to first rescue analgesia, opioid consumption, postoperative nausea and vomiting (PONV) score, and complications, and to determine which one is more effective.

DETAILED DESCRIPTION:
VATS (Video-Assisted Thoracoscopic Surgery) is based on the principle of performing surgical procedures through two 2-3 cm skin incisions into the thorax with instruments inserted through an endocamera placed in the thoracic cavity, and the images reflected on a monitor. The procedure is carried out in operating room conditions under general anesthesia. Collapsing the lung on the same side during the procedure allows exploration of the thoracic cavity and facilitates the free movement of surgical instruments within the cavity. Patients are placed in the lateral decubitus position on the operating table, and preparations are made for posterolateral thoracotomy in case the method proves insufficient or complications arise. A 2 cm skin incision is made at the 7th or 8th intercostal space (ICS) on the mid-axillary line. After blunt dissections, muscles are passed through, and the parietal pleura is opened. The lung collapses with the developing pneumothorax. Digital palpation checks for pleural adhesions, and the endocamera is inserted into the thorax. After exploration, the locations for the insertion of surgical instruments are determined for the other ports. Depending on the lesion's localization, two or more ports are opened. VATS has recently been considered a standard surgical procedure for lung surgery. Compared to open thoracotomy, the advantages of VATS surgery include rapid recovery, shorter hospitalization, and a lower risk of complications. Although VATS surgery is less painful than thoracotomy, especially in the first hours after VATS surgery, severe acute postoperative pain can occur. Thoracic epidural analgesia (TEA), the gold standard for post-thoracotomy analgesia, is also used for VATS postoperative analgesia. However, due to differences in surgical technique and trauma between open surgery and VATS, there is a debate about what the gold standard for post-VATS analgesia should be. Especially due to the difficulty of TEA application and the side effect profile of hypotension, urinary retention, or nausea/vomiting, there is support for the application of less invasive analgesic techniques for minimally invasive surgical procedures. Postoperative pain in patients undergoing VATS is observed, although not as severe as post-thoracotomy pain. This, like in thoracotomy, affects postoperative pulmonary complications and the length of hospitalization for patients. If postoperative acute pain is not adequately treated, it can lead to chronic pain in the long run. In recent years, regional anesthesia techniques are frequently applied to patients for pain management, in addition to general anesthesia (GA). TPVB, ESPB, and SAPB are among the commonly used regional anesthesia techniques in thoracic surgery. GA is the basic anesthesia method for thoracic surgery. However, GA can only inhibit the cortical limbic system or the projection system of the hypothalamic cortex. It cannot completely block the transmission of peripheral noxious stimuli to the central nervous system or effectively prevent the intraoperative stress response. Consequently, the intensive use of opioid analgesics accompanies GA. The intense use of opioids leads to delayed extubation, respiratory depression, nausea, and vomiting. Adding peripheral blocks such as TPVB and SPSIPB is expected to provide preemptive analgesia, resulting in more stable hemodynamics and less intraoperative opioid use. TPVB has long been a primary regional technique for VATS surgery in the literature. In addition, SPSIPB performed under ultrasound guidance, defined by Tulgar and colleagues in 2023, has become a routine interfacial plane block applied as needed. It is based on the injection above the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in conditions such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. The SPS muscle is located at the C7-T2 level, attaching to the lateral edges of the second and fifth ribs. It is innervated by the lower cervical and upper intercostal nerves. Analgesia is provided by blocking these nerves with SPSIPB. In a cadaver study conducted by Tulgar and colleagues, the spread of SPSIPB was observed as staining in a speckled pattern only on the surface fascia of the trapezius muscle at 7-10 intercostal levels on the left side, with no staining on the right side. Clear staining was observed deep in the trapezius muscle on both sides. The deep and superficial parts of the rhomboid major were clearly stained, while only the deep part of the rhomboid minor was stained. It was emphasized that SPSIPB provides successful analgesia in procedures involving the thoracic region, such as chronic myofascial pain, breast surgery, thoracic surgery, and shoulder surgery.

Materials and Methods:

This study is a prospective, randomized, double-blind observational trial. A minimum of 70 patients, aged between 18 and 65, with a body mass index (BMI) <35, undergoing VATS surgery at the Chest Surgery Service of Hitit University Faculty of Medicine Erol Olçok Training and Research Hospital, and classified under the American Society of Anesthesiologists (ASA) physical classification 1-2-3, who have read and accepted the voluntary informed consent form, will be included. Patients will be randomly assigned to two groups using a computer-based method. The study will be blinded for patients, surgeons, and those monitoring postoperative pain. Group T (n=35) will consist of patients receiving TPVB, and Group S (n=35) will include patients receiving SPSIPB.

Exclusion criteria:

Patients unwilling to participate in the study, those with BMI >35, ASA 4-5 classification, inability to score pain using the Visual analog score (VAS) system, allergies to the local anesthetic and specified analgesic drugs, pregnant or breastfeeding women, patients under 18 or over 65 years old, those with uncontrolled anxiety, alcohol or drug dependence, neuromuscular or peripheral nerve diseases, high-dose opioid use 3 days before surgery, widespread chronic pain, diabetes mellitus, hepatic and renal insufficiency, coagulation disorders, and patients using anticoagulant drugs, as well as those with infections at the site of peripheral block needle entry, a history of abdominal surgery or trauma, inability to communicate in Turkish, technical problems while using patient-controlled analgesia (PCA) during surgery, and patients for whom surgery needs to be terminated before completion and those for whom postoperative extubation is not planned will be excluded from the study.

Method:

Patients will be provided with the necessary information about the procedure, and written consent will be obtained. Included patients will be randomly assigned to either Group T or Group S according to a computerized randomization table created by a non-participating researcher. Each patient will be assigned a random code for blinding, sealed in envelopes. The anesthetist in the operating room will receive the relevant sealed envelope indicating the block to be performed for each randomized patient. Patients, surgeons, and those monitoring postoperative pain will be blinded to the patient's group information. Patients will be taken to the operating room, where standard anesthesia monitoring will be applied. (non-invasive arterial blood pressure measurement, heart rate, electrocardiography, peripheral oxygen saturation measurement). A 20 G catheter will be placed for intravenous access in the patient. The time of anesthesia initiation will be recorded. For premedication, 0.03 mg/kg midazolam will be administered to the patients, and after preoxygenation, anesthesia induction will be performed with 2 mg/kg propofol and 1 mcg/kg fentanyl. After the administration of 0.6 mg/kg rocuronium bromide IV and achieving muscle relaxation, intubation will be performed with a double-lumen endotracheal tube. Mechanical ventilation will be provided with pressure-controlled mode targeting an end-tidal CO2 value of 35-40 mmHg. During anesthesia maintenance, O2/air mixture (FiO2: 0.40), sevoflurane (minimum alveolar concentration 0.8-1), and IV remifentanil infusion will be used. Remifentanil infusion will be planned to maintain the patient's mean arterial blood pressure within 20% of the baseline value. The patient's intraoperative vital signs will be monitored as per routine anesthesia protocol. As an intraoperative antiemetic, 4 mg ondansetron IV will be administered. Thirty minutes before the end of the surgical procedure, 1 g of paracetamol infusion and 1 mg/kg contramal IV infusion will be administered to all patients for analgesic purposes. After the completion of the surgery, while maintaining the depth of anesthesia, the regional anesthesia technique will be applied. All block procedures will be performed under sterile conditions. The end time of the surgical procedure, the end time of anesthesia, the time of block administration, and the time of anesthesia termination will be recorded.

SPSIPB Technique:

The SPSIPB block, which follows the guidelines we routinely use, will be performed after the completion of the surgical procedure and before the patient wakes up. A high-frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The procedure will be performed with the patient in a lateral decubitus position. After gently shifting the scapula laterally, the US probe will be held sagittally at the upper corner of the scapula spine, visualizing the 3rd rib and the serratus posterior superior muscle. An in-plane technique will be used. The block needle will be advanced cranio-caudally between the serratus posterior superior and the 3rd rib. Block placement will be confirmed by injecting 5 ml of saline between the rib and muscle. After confirming the block placement, 30 ml of 0.25% concentration marcain (bupivacaine) will be used.

TPVB Technique:

The US probe (11-12 MHz, Vivid Q) will be placed 2-3 cm lateral to the T5 spinous process. After visualizing the transverse process, the paravertebral area, internal intercostal membrane, paravertebral space, and pleura, the needle will be advanced to the paravertebral space using an in-plane technique. Hydrodissection with 5 ml of saline and pleural depression will be performed in this area. After confirming the accuracy of the site, 30 ml of 0.25% bupivacaine will be injected into this area.

After completing the designated block procedure, neuromuscular blockade will be reversed with 4 mg/kg sugammadex under 80% O2 ventilation. After confirming spontaneous eye opening, the endotracheal tube will be removed, and patients will be transferred to the intensive care unit for observation and close monitoring. Postoperative pain monitoring, blinded to the patient's group information, will be performed by an

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 70 patients who will undergo VATS surgery,
* American Society of Anesthesiologists (ASA) physical classification 1-2-3,
* Aged between 18-65,
* Who have read and accepted the voluntary informed consent form,
* Body mass index (BMI) of <35.

Exclusion Criteria:

* Patients who refuse to participate in the study,
* BMI >35,
* ASA physical classifications 4-5,
* Patients unable to perform pain scoring using the NRS system,
* Those allergic to the administered local anesthetic and designated analgesic medication, individuals declaring pregnancy or lactation,
* Patients under 18 or over 65 years of age,
* Uncontrollable anxiety,
* Alcohol and drug addiction,
* Neuromuscular and peripheral nerve diseases,
* Using high doses of opioid medication three days before surgery,
* Widespread chronic pain,
* Diabetes mellitus,
* Hepatic and renal insufficiency,
* Coagulation disorders,
* Using anticoagulant drugs,
* Infection at the site of peripheral block needle insertion,
* History of abdominal surgery or trauma,
* Unable to communicate in Turkish,
* Patients experiencing technical problems while using patient-controlled analgesia,
* Patients for whom the surgical procedure needs to be terminated for any reason before completion, as well as those for whom postoperative extubation is not planned, will not be accepted into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Postoperatative Pain | 24 hours
  Evaluation of patients' post-operative pain levels

CONTACTS AND LOCATIONS:
Overall Officials: Guvenc Dogan, MD, Study Chair — Hitit Universirty
Locations (1):
- Hitit university, Çorum, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
not necessary